CLINICAL TRIAL: NCT04311359
Title: A Pharmacovigilance Study of Brain Oedema in the Food and Drug Administration Adverse Event Reporting System Using Data Mining Algorithms
Brief Title: A Pharmacovigilance Study of Brain Oedema
Status: Completed | Type: Observational
Sponsor: University of Peshawar (Other)
Responsible Party: Principal Investigator, Mohammad Ismail, Assistant Professor, Department of Pharmacy, University of Peshawar
Other Study IDs: PV-BO
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Brain Edema; Brain Edema Caused by Drugs
MeSH Terms: conditions — Brain Edema | interventions — Drugs, Generic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Group/Cohort: Brain Oedema induced by drugs reported to the FAERS database from inception till first quarter of 2019
  Interventions: Drug: Drugs, Generic

INTERVENTIONS:
Drug: Drugs, Generic — All drugs having 19 or more Brain Oedema cases reported to the FAERS database

SUMMARY:
Literature reports the development of brain oedema following the use of certain drugs. Therefore, this study aims to present a comprehensive disproportionality analysis of brain oedema cases reported to the Food and Drug Administration Adverse Event Reporting System (FAERS).

DETAILED DESCRIPTION:
Brain oedema is a serious neurological condition, as it possesses a significant impact on the functional abilities of an individual by causing irreversible brain damage and potentiates the risk of mortality. Apart from a number of medical conditions causing brain oedema, evidence suggests the association of various drugs with brain oedema. Therefore, this study aims to provide a comprehensive disproportionality analysis of the drug-induced brain oedema reports in the FAERS database.

ELIGIBILITY:
Inclusion Criteria:

* Brain Oedema cases reported in the FAERS database till 31/03/2019
* Adverse event reported was included using the MedDRA term: Brain Oedema

Exclusion Criteria:

* Drugs with less than 19 brain oedema reports

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presented with brain oedema treated for any disease
Sampling Method: Non-Probability Sample
Enrollment: 9524 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Identification of drugs associated with Brain Oedema | Cases reported to the FAERS database since inception till 31/03/2019
  The search includes MedDRA (v-22) Preferred Term, "Brain Oedema (MedDRA code: 10048962) for the identification of all Brain Oedema case reports and drugs.
Detection of signals of Brain Oedema | Cases reported to the FAERS database since inception till 31/03/2019
  Signal detection using disproportionality analysis

SECONDARY OUTCOMES:
Stratification of new signals with respect to age | Cases reported to the FAERS database since inception till 31/03/2019
Stratification of new signals with respect to gender | Cases reported to the FAERS database since inception till 31/03/2019
Trends of Brain Oedema reports in FAERS database | Cases reported to the FAERS database since inception till 31/03/2019
Trends of Brain Oedema reports in Google searches | Cases reported to the FAERS database since inception till 31/03/2019
Description of the population of patients having Brain Oedema | Cases reported to the FAERS database since inception till 31/03/2019

CONTACTS AND LOCATIONS:
Locations (1):
- University of Peshawar, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided